CLINICAL TRIAL: NCT04334278
Title: Development of a Mind Body Program for Obese Knee Osteoarthritis Patients With Comorbid Depression: Does a Mind Body Program Reduce Osteoarthritis Pain?
Brief Title: Development of a Mind Body Program for Obese Knee Osteoarthritis Patients With Comorbid Depression
Acronym: GetHealthy-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Caitlin Conley, Assistant Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67336; 5R34AT010370-03 (NIH)
Record Dates: First submitted 2020-03-30; First posted 2020-04-06 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis; Obesity; Depression
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GetHealthy-OA (Experimental): The GetHealthy-OA is an 6-week group mind body program with efficacy in improving depression, physical function and aiding in weight loss, that has been adapted for the unique needs of patients with knee osteoarthritis, depression and obesity. The GetHealthy-OA will be delivered by secure telehealth.
  Interventions: Behavioral: GetHealthy-OA
- Health Enhancement Program (Active Comparator): The Health Enhancement Program is a chronic pain-specific program adapted for the specific needs of patients with knee osteoarthritis. It is an 6-week group mind body program that will be delivered via secure telehealth. To control for in between session practice, participants will receive an mp3 recording and informational handout to complete after each session.
  Interventions: Behavioral: Health Enhancement Program

INTERVENTIONS:
Behavioral: GetHealthy-OA — The GetHealthy-OA is an 6-week group mind body program with efficacy in improving depression, physical function and aiding in weight loss, that has been adapted for the unique needs of patients with knee osteoarthritis, depression and obesity. The GetHealthy-OA will be delivered by secure telehealth.
  Arms: GetHealthy-OA
Behavioral: Health Enhancement Program — The Health Enhancement Program is a chronic pain-specific program adapted for the specific needs of patients with knee osteoarthritis. It is an 6-week group mind body program that will be delivered via secure telehealth.
  Arms: Health Enhancement Program

SUMMARY:
Knee osteoarthritis (OA) is the most common joint disorder in the U.S. and a leading cause of disability. Depression and obesity are highly comorbid among knee osteoarthritis patients, and the combination of obesity and depression is associated with decreased physical activity, higher pain and disability, and more rapid cartilage degradation. Depression, obesity and osteoarthritis exacerbate one another and share a common pathophysiology involving systemic inflammation and pro-inflammatory cytokines, reflecting a complex mind-body interaction. Current treatments for knee osteoarthritis offer little to no benefit over placebo, and do not emphasize mind-body practices or physical activity to target the underlying pathophysiology. Mind-body interventions to lessen depressive symptoms and increase physical activity offer the ability to target biological, mechanical and psychological mechanisms of osteoarthritis progression in this high-risk subset. The long-term goals are to evaluate the mechanisms by which the Relaxation Response Resiliency Program (3RP) delivered via telehealth, and adapted for patients with depression, obesity and knee OA (GetHealthy-OA) promotes increases in physical activity and improved subjective and objective aspects of knee health. The overarching hypothesis is that the synergistic interaction between mindfulness, adaptive thinking, positive psychology and healthy living skills of the GetHealthy-OA will reduce pro-inflammatory cytokine expression while also promoting optimal mechanical loading of the cartilage thereby slowing the progression of symptomatic knee osteoarthritis. This study aims to adapt the 3RP for the needs of knee osteoarthritis patients with depression and obesity with a focus of increasing physical activity, and iteratively establish the feasibility, credibility and acceptability of the programs and research procedures.

DETAILED DESCRIPTION:
The conceptual model of adaptation of the general 3RP to obese osteoarthritis patients with depression that specifically target improved function through combining mind body skills with physical activity, and recommendations of multimodal programs to improve outcomes in chronic pain clinical trials. Adaptations of the multimodal general 3RP will be done consistent with theoretical models of the fear-avoidance model of pain, cognitive model of pain and depression, acceptance and commitment therapy, mindfulness, and positive psychology. The goal is to help patients engage in activities that are meaningful and mapped to each individual's level of functioning and life circumstance through the use of quota-based pacing through adaptation of skills to directly address improved mood, healthy lifestyle (sleep, diet), correction of knee osteoarthritis misconceptions, and use of relaxation response elicitation and positive psychology skills to promote awareness and calm during activities, even when these are painful.

The guiding hypothesis is that the synergistic interaction between mindfulness, adaptive thinking, positive psychology, physical activity and healthy living skills of the GetHealthy-OA reduces pro-inflammatory cytokine expression while also promoting optimal mechanical loading of the cartilage thus slowing the progression of symptomatic knee OA. In this project the 3RP will be iteratively adapted for the needs of knee osteoarthritis patients with depression and obesity with a focus on gradual increases in physical activity measured with accelerometers and establish feasibility markers for the program and procedures. A pilot randomized controlled trial of the GetHealthy-OA versus a time- and attention-matched health enhancement control will be performed to assess the feasibility of recruitment procedures, feasibility and acceptability of the GetHealthy-OA and control, and data collection procedures by group.

A pilot randomized controlled trial (N=60 participants) of the GetHealthy-OA with a time and attention matched health enhancement control will be performed. The end goal of the pilot RCT is not to assess the efficacy of the GetHealthy-OA but rather to assess the feasibility of recruitment procedures (screening, eligibility, enrollment rates), feasibility and acceptability of the GetHealthy-OA and control intervention (adherence, retention, fidelity, satisfaction, group telehealth delivery, and data collection procedures by group (adherence, satisfaction, blood and urine biomarker data).

A single blind pilot feasibility randomized controlled trial with a time, dose and attention matched health enhancement control will be conducted (N=60; approximately 5 GetHealthy-OA groups and 5 control, 6-8 per group). Participants will be randomized in a 1:1 design using a randomization scheme developed by the statistician. Research procedures will be identical for patients in GetHealthy-OA and control. The study will yield information on how participants might engage differently with the intervention and control, definitive information on feasibility and acceptability and signal of improvement in the intervention before investment of resources in the full randomized controlled trial.

The GetHealthy-OA refined based on exit interviews and surveys. The control group will have the same format as the GetHealthy-OA, and the control group follows the format of the Health Enhancement Program. A pain specific adaptation of this program for chronic pain exists. This program will be adapted for the specific needs of patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients (BMI > 30 kg/m2)
* Idiopathic knee OA per the American College of Rheumatology classification with mild to moderate radiographic changes (Kellgren/Lawrence grade 2 or 3)
* Current elevated depressive symptoms (PHQ-9 > 9)
* Age 45 or older
* Free of concurrent psychotropics for < 2 weeks prior to initiation of treatment or on stable doses for > 6 weeks
* Access to a computer/smart phone with internet access
* Willingness to comply with the study protocol and assessments
* Cleared by a medical doctor to participate

Exclusion Criteria:

* Any disorder requiring the use of systemic corticosteroids
* Rheumatoid arthritis
* History of cancer within 5 years of screening
* Unable to walk/wheelchair-bound
* Prior surgical fixation of a femur or tibia fracture
* Taking high doses of opioid pain medication (50 milligrams of morphine equivalent)
* Diagnosis of a medical illness expected to worsen in the next 6 months (e.g., malignancy)
* Active suicidal ideation or past-year psychiatric hospitalization
* Non-English speaking
* Current severe depression symptoms (PHQ-9 > 19)
* Lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder
* Current substance abuse or dependence
* Substance use disorder within the past 6 months
* Practice of yoga/meditation, or other mind body techniques that elicit the relaxation response, once per week for 45 min or more within the last 3 months
* Engagement in regular moderate or vigorous physical exercise for >30 min daily

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Conley, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - UK Healthcare at Turfland, Lexington, Kentucky
  - UK HealthCare Joint Reconstruction and Replacement, Lexington, Kentucky

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 66 patients were enrolled. However, 15 participants were excluded prior to randomization/group assignment because they were lost to follow-up when scheduling baseline testing.
Period: Overall Study
Arm/Group | GetHealthy-OA | Health Enhancement Program
Started | 28 | 23
Completed | 24 | 18
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GetHealthy-OA | Health Enhancement Program | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (6) | 56 (8) | 55 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 28 | 22 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 19 | 15 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 23 | 51

OUTCOME MEASURES:

1. Primary Outcome: Treatment Adherence
Description: Number of patients that attend a minimum of 4 of 6 weekly sessions
Time Frame: 6-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GetHealthy-OA | Health Enhancement Program
Number analyzed (Participants) | 28 | 23
Participants | 24 | 18

2. Secondary Outcome: Accelerometer Compliance
Description: Number of days participants wore the Accelerometers at least 8 hours per day
Time Frame: Baseline, 6 weeks
Measure: Mean (Full Range); unit: days
Arm/Group | GetHealthy-OA | Health Enhancement Program
Number analyzed (Participants) | 28 | 23
days
  Baseline | 6 [0 to 7] | 6 [1 to 7]
  6-weeks | 3 [0 to 7] | 4 [0 to 7]

3. Secondary Outcome: Number of Missing Specimens
Description: Number of missing blood or urine specimens per patient
Time Frame: Baseline, 6 weeks
Measure: Count of Units; unit: Specimens
Units Other Than Participants: Specimens
Arm/Group | GetHealthy-OA | Health Enhancement Program
Number analyzed (Participants) | 28 | 23
Number analyzed (Specimens) | 56 | 46
Specimens
  Baseline - blood | 1 | 0
  6-weeks - blood | 7 | 6
  Baseline - urine | 6 | 5
  6-weeks - urine | 12 | 17

4. Secondary Outcome: Daily Practice Adherence
Description: Number of patients that completed daily practice at least 4 days per week
Time Frame: 6 weeks
Population: As part of the intervention the GetHealthy-OA group was the only group to have homework. The Health Enhancement Program didn't have any recorded homework, which is why there is daily practice adherence listed for the Health Enhancement Program.
Measure: Count of Participants; unit: Participants
Arm/Group | GetHealthy-OA
Number analyzed (Participants) | 28
Participants | 18

ADVERSE EVENTS:
Time Frame: Data was collected during an 8-week period (6-weeks for the program, 1-week for pre-testing, and 1-week for post-testing)
Arm/Group | GetHealthy-OA | Health Enhancement Program
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/23
Other Adverse Events (participants affected / at risk) | 0/28 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT04334278/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT04334278/ICF_000.pdf